CLINICAL TRIAL: NCT06858592
Title: Osteopathic Manipulative Techniques in Collegiate Dancers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Collaborators: University of Louisiana Monroe (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2024-181
Record Dates: First submitted 2025-02-24; First posted 2025-03-05 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-02

CONDITIONS: Osteopathic Manipulative Treatment (OMT); Dance Therapy
Keywords: Dance; Osteopathic Manipulative Treatment (OMT); Mental Health; Athletic Identity
MeSH Terms: conditions — Psychological Well-Being | interventions — Manipulation, Osteopathic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment Population (Experimental): This pilot study will collect data from, diagnose, treat, and reassess dancers on the ULM dance team. They will be asked to complete multiple questionnaires and a survey to determine their medical history, dance background, and mental health. The Multidimensional Pain Questionnaire in Professional Dance (MPQDA) will be used to collect dancer demographics, history, and performance-related pain levels. The Dance Functional Outcome Survey (DFOS) will collect data on the dancers' areas of pain and perceived movement quality and function while performing. Then, the dancer will be treated for 15 minutes using OMT by the osteopathic medical student and supervising physician beginning with the area of greatest restriction within the lower body, including the lumbar spine, hips, knees, ankles, and feet. Following diagnosis and treatment, dancers will attend a dance practice, and be re-evaluated immediately afterward. After 24 hours, dancers will be evaluated again with the force plate.
  Interventions: Procedure: Osteopathic Manipulative Treatment (OMT)

INTERVENTIONS:
Procedure: Osteopathic Manipulative Treatment (OMT) — Dancers will then individually be screened for somatic dysfunctions (SD) by a physician and VCOM OMS-III student doctor under their direct supervision. OMS-III student investigators will receive training and be assessed on their abilities before performing OMT on subjects. This will take place at the dancers' place of practice in a private area equipped with an OMM table. The areas to be screened include the lumbar spine, hips, knees, ankles, and feet. All diagnoses in these areas will be documented with specific notation for the area of greatest restriction on paper. After making a diagnosis or multiple diagnoses, the dancer will be treated utilizing OMT for 15 minutes starting with the area of greatest restriction in the lower body by the OMS-III student doctor under direct supervision of a physician, should an adverse event take place. The type of treatment(s) used will be at the discretion of the supervising physician and the VCOM student doctor. They may use any OMT technique, exc

SUMMARY:
The goal of this study is to determine how these techniques affect pain levels, movement quality, and balance. Osteopathic Manipulative Techniques, or OMT, is a type of treatment used to treat problems in the bones, muscles, tissues, and joints. The investigators would like to ask the participants to fill out a few questionnaires about their personal history, dance background, pain levels, and movement quality. All participant responses will be completely anonymous, and participants are allowed to refuse to answer any part of the survey. The investigators would also ask participants to complete a balance assessment, which will involve standing on a force plate with their eyes open and closed for 30 seconds each. The initial survey and questionnaires, balance assessment, OMT, and post-practice survey are expected to take about 60 minutes. Each additional survey given after 24-hours and one week will take about 20 minutes each. The follow-up balance test after one week is expected to take less than 5 minutes. Participation in this study would be immensely valuable for us to learn more about the benefits of treating dancers with osteopathic manipulative medicine.

DETAILED DESCRIPTION:
Many dancers base their identities and self-worth on being able to train, rehearse, and perform. Because of this, dancers are more likely to ignore any pain or discomfort and continue dancing, despite the risk of worsening pain or injuries. Injuries are very common in dancers due to repetitive motions, overuse of muscles and joints, improper technique, acute injuries, or energy balance deficits. The most common areas of pain and injury seen in dancers include the hips, knees, ankles, feet, and lumbar spine. While many current treatments are available for dance-related pain and injuries, many of them involve rest and time off from dancing, which many dancers are not willing to do. Although Osteopathic Manipulative Treatment (OMT) is not a substitute for rehabilitation and other treatments necessary for injuries, it may enhance their recovery time and prevent future injuries. This study aims to examine the significance of utilizing OMT to decrease dancers' performance-related pain, increase dancers' movement quality, and increase dancers' balance. OMT is the manipulation of the musculoskeletal system to assist the body in healing and strengthening itself while encouraging resistance to future stressors. Athletes, such as dancers, may find OMT beneficial for decreasing their pain, improving their range of motion, and preventing future injuries. Other athletes have reported satisfaction with OMT modalities in decreasing their injury-related pain and stress, decreasing their need for pain medications, and enhancing their recovery and return to activity. The purpose of this pilot study is to assess dancers' perceived performance-related pain, movement quality, and balance before and after OMT in the regions of the lumbar spine, hips, knees, ankles, and/or feet. Additionally, this study will collect data on the dancers' self-identity in relation to their role as athletes and potential risk factors for disordered eating. Future goals include conducting a larger study to treat and prevent dance-related injuries. Dancers from the University of Louisiana Monroe (ULM) dance team will be recruited to participate in this study. All dancers who choose to participate will be in the experimental group, there will not be a control group. Dancers will complete a survey and questionnaires to provide demographic information, their medical history, dance background, attitudes towards eating, ways in which they identify as an athlete, performance-related pain levels, and perceived movement quality and function while dancing. Dancers will also complete two 30-second balance tests with their eyes open and closed. Following completion of these forms and tests, dancers will be screened for somatic dysfunction(s) and treated appropriately by a medical student from the Edward Via College of Osteopathic Medicine - Louisiana (VCOM) and a supervising physician. After treatment, dancers will attend their practice as normal. Following this, study participants will be re-evaluated immediately after the dance practice, 24 hours later, and one week later. The results of this study may be utilized to write a paper, create a poster presentation, and support a larger study in the future. Significant results would be beneficial in the field of sports medicine to help guide appropriate treatment in dancers and provide more treatment options to allow them to continue dancing.

ELIGIBILITY:
Inclusion Criteria:

* Members of the ULM dance team (HawkLine)

Exclusion Criteria:

* Non-competitive members of the team, those injured and those that opt out of the study.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-02-22 (Actual); Study Completion 2025-02-22 (Actual)

PRIMARY OUTCOMES:
Changes in perceived pain after Osteopathic Manipulative Treatment (OMT) | 7 days
  The Multidimensional Pain Questionnaire in Professional Dance (MPQDA) will be used to collect dancer demographics, history, and performance-related pain levels. The questionnaire includes the following blocks (questions contents are in parentheses):prevalence and localizations; subjective sensation of pain; temporal course of pain. On a four-point ordinal scale from 'not' (= 0) to 'very' (= 3), accompanying symptoms (tension, redness, swelling, warming, restrictions of mobility and resilience) are asked.
Changes in balance after Osteopathic Manipulative Treatment (OMT) | 7 days
  This pilot study will utilize the IsoBALANCE® force plate and scoring system to balance in collegiate dancers before and after receiving OMT. Distance in CM traveled along X and Y axis will be measured during 2 30-second bouts: the first with eyes open and the second with eyes closed. A radius of movement from center (in cm) will also be calculated.
Changes in performance after Osteopathic Manipulative Treatment (OMT) | 7 days
  The Dance Functional Outcome Survey (DFOS) will collect data on the dancers' areas of perceived movement quality and function while performing. 14 questions in the areas of ADL and dance/technique specific "requiring answers of agreement or disagreement to a statement" Max of 40 points; 1 general dance performance grade question (0-100 scale); and Technique section: Max 50 points. Higher score reflects higher function.
Changes in performance after Osteopathic Manipulative Treatment (OMT) | 7 days
  Screening 6 from Athlete's Form #2 on the International Olympic Committee Sport Mental Health Assessment Tool 1 (SMHAT-1) will be used to screen for eating habits and attitudes toward food, eating, weight, and body image that may identify risk factors of disordered eating. The 9-item screen asks about food attitudes over the previous 14 day period. It is scored on a 3 to Zero scale (3=always, 0=sometimes/rarely/never) with higher scores indicating more risk for disordered eating. Topics included guilt after eating; desire to be thinner; satisfaction with body shape; trying to lose weight; avoidance of disappointing parents.
Changes in performance after Osteopathic Manipulative Treatment (OMT) | 7 days
  The Athletic Identity Measurement Scale (AIMS) measures the degree to which an individual identifies with the athlete role. The AIMS is a 10-item self-report questionnaire that was developed to assess domain-specific self-identification as an athlete. The original 10-item AIMS version produced a more has been used in investigations of a wide variety of sport-related phenomena from its 3 sub-scales: social identity, exclusivity, and negative affectivity. For this study, the participants will complete the 10-item version. 8 of the items are worded positively; 2 are worded negatively (inversely scored) using a 1 to 7 Likert scale (Strongly disagree to Strongly agree).

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie N Aldret, DO, CAQSM, FAOASM, Principal Investigator — Edward Via College of Osteopathic Medicine
Locations (1):
- Edward Via College of Osteopathic Medicine, Monroe, Louisiana, United States

IPD SHARING:
Plan to Share IPD: Undecided
To protect the anonymity of the study subjects.

REFERENCES:
- [Background] Bowling A. Injuries to dancers: prevalence, treatment, and perceptions of causes. BMJ. 1989 Mar 18;298(6675):731-4. doi: 10.1136/bmj.298.6675.731. PMID 2496824
- [Background] Werber B. Dance medicine of the foot and ankle: a review. Clin Podiatr Med Surg. 2011 Jan;28(1):137-54. doi: 10.1016/j.cpm.2010.10.005. PMID 21276523
- [Background] Opdam KTM, van Loon J, Zwiers R, Kuijer PPFM, van Dijk CN. Corticosteroid Injections in Posterior Ankle Impingement Syndrome: A Survey of Professional and Elite Student Ballet Dancers. J Dance Med Sci. 2021 Mar 15;25(1):24-29. doi: 10.12678/1089-313X.031521d. PMID 33706852
- [Background] 10. Teitz, C. C. (2000). Hip and knee injuries in dancers. Journal of Dance Medicine & Science, 4(1), 23-29. https://doi.org/10.1177/1089313x0000400105
- [Background] Sammarco GJ. Diagnosis and treatment in dancers. Clin Orthop Relat Res. 1984 Jul-Aug;(187):176-87. PMID 6146421
- [Background] 7. Mainwaring, L. M., Krasnow, D., & Kerr, G. (2001). And the dance goes on: Psychological impact of injury. Journal of Dance Medicine & Science, 5(4), 105-115. https://doi.org/10.1177/1089313x0100500402
- [Background] Gunnar Brolinson P, McGinley SM, Kerger S. Osteopathic manipulative medicine and the athlete. Curr Sports Med Rep. 2008 Feb;7(1):49-56. doi: 10.1097/01.CSMR.0000308664.13278.a7. PMID 18296946
- [Background] Ofei-Dodoo S, Black JL, Kirkover MA, Lisenby CB, Porter AST, Cleland PM. Collegiate Athletes' Perceptions of Osteopathic Manipulative Treatment. Kans J Med. 2020 Jun 25;13:147-151. eCollection 2020. PMID 32612747
- [Background] Shah S, Weiss DS, Burchette RJ. Injuries in professional modern dancers: incidence, risk factors, and management. J Dance Med Sci. 2012 Mar;16(1):17-25. PMID 22390950
- [Background] 2. Malkogeorgos, A., Mavrovouniotis, F., Zaggelidis, G., & Ciucurel, C. (2011). Common dance related musculoskeletal injuries. Journal of Physical Education and Sport, 11(3).
- [Background] Benardot D. Nutritional Concerns for the Artistic Athlete. Phys Med Rehabil Clin N Am. 2021 Feb;32(1):51-64. doi: 10.1016/j.pmr.2020.09.008. Epub 2020 Oct 29. PMID 33198898